CLINICAL TRIAL: NCT01410812
Title: Tying Devices as a Means of Increasing Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 813970; NCT01421329 (obsolete NCT alias)
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Interest in exercising more

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Suggested Tying (Experimental): Receive same treatments as control group, but instead of receiving cash they receive 4 iTunes audio novels for their own iPods. Further, they are prompted to try to listen to those novels only when exercising at the gym in order to increase their attendance.
  Interventions: Behavioral: Suggested Tying Intervention
- Forced Tying (Experimental): Receives same treatment as the control group. However, in addition to receiving the cash, they also receive 4 iTunes audio novels for a loaned iPod that they will only have access to at the gym. They are told they may only listen to these novels only when at the gym in order to increase their attendance.
  Interventions: Behavioral: Forced Tying Intervention
- Control (Experimental): Control group of participants who do not receive any intervention but are weighed at the beginning and end of a 10 week period and receive weekly emails asking them about their exercise. They also receive the equivalent cash value of 4 iTunes audio novels
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Control — Receive weekly emails asking participants about their exercise and receive cash.
  Arms: Control
Behavioral: Suggested Tying Intervention — Participants receive 4 iTunes audio novels for their own iPods to listen to only at the gym
  Arms: Suggested Tying
Behavioral: Forced Tying Intervention — Participants receive cash and also 4 iTunes audio novels for a loaned iPod accessible only at the gym to listen to only at the gym.
  Arms: Forced Tying

SUMMARY:
The investigators propose that healthy behaviors such as exercise could be increased through the use of tying devices - mechanisms that force a coupling of addictive activities (listening to the next chapter of a page-turner novel) with engagement in a healthy behavior (exercise).

DETAILED DESCRIPTION:
The study will test the effect of the following treatments as a means of increasing gym attendance over 10 weeks: 1. Participants receive access to 4 iTunes audio novels on their own iPods and prompted to listen to those novels only when exercising at the gym; 2: Participants receive 4 iTunes audio novels for a loaned iPod that they will only have access to at the gym; 3: Participants receive weekly emails asking them about their exercise.

ELIGIBILITY:
Inclusion Criteria:

* Stable health as determined by the screening of their medical history
* Own an iPod
* An interest in exercising more regularly
* Belong to the Pottruck Gym at University of Pennsylvania
* Interested in exercising more through the use of aerobic exercise machines

Exclusion Criteria:

* Recent myocardial infraction
* congestive heart failure
* uncontrolled hypertension
* self-report of 6 or more alcoholic beverages per day or use of any illicit drugs
* bulimia nervosa or related behaviors
* diabetes medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L. Milkman, Ph.D., Principal Investigator — University of Pennsylvania; Julia A Minson, Principal Investigator — University of Pennsylvania; Kevin G.M. Volpp, MD, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suggested Tying | Forced Tying | Control
Started | 75 | 75 | 76
Completed | 75 | 75 | 76
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suggested Tying | Forced Tying | Control | Total
Number analyzed (Participants) | 75 | 75 | 76 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 75 | 75 | 76 | 226
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 48 | 149
  Male | 25 | 24 | 28 | 77

OUTCOME MEASURES:

1. Primary Outcome: Average Weekly Gym Attendance From Baseline to Week 9
Time Frame: 9 weeks
Measure: Mean (95% Confidence Interval); unit: Average Weekly Gym Attendance
Arm/Group | Suggested Tying | Forced Tying | Control
Number analyzed (Participants) | 75 | 75 | 76
Average Weekly Gym Attendance | 1.21 [1.05 to 1.37] | 1.42 [1.25 to 1.59] | 0.94 [0.78 to 1.10]

2. Secondary Outcome: Dollar Amount Participants Would Pay for Enrollment
Description: Willingness to pay is measured as the dollar amount a participant would pay to be enrolled in a program such as the treatment. Participant who would pay more are said to be more willing to pay, as opposed to those who would pay less or not at all.
Time Frame: 9 weeks
Population: Some of the participants failed to respond for this outcome measure.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Suggested Tying | Forced Tying | Control
Number analyzed (Participants) | 71 | 69 | 71
Dollars | 4.77 (7.24) | 6.01 (8.31) | 9.87 (14.55)

ADVERSE EVENTS:
Arm/Group | Suggested Tying | Forced Tying | Control
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75 | 0/76
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes